CLINICAL TRIAL: NCT01298700
Title: A 2-year, Multicenter, Double-masked, Randomized, Parallel Study of the Safety of LUMIGAN® 0.1 mg/mL Compared With LUMIGAN® 0.3 mg/mL in Patients With Glaucoma or Ocular Hypertension
Brief Title: Long-Term Safety of Bimatoprost Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192024-054; 2010-023917-68 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-12

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bimatoprost 0.01% Ophthalmic Solution (Experimental): One drop of bimatoprost 0.01% ophthalmic solution instilled to each eye, once daily in the evening for 2 years.
  Interventions: Drug: bimatoprost 0.01% ophthalmic solution
- Bimatoprost 0.03% Ophthalmic Solution (Active Comparator): One drop of bimatoprost 0.03% ophthalmic solution instilled to each eye, once daily in the evening for 2 years.
  Interventions: Drug: bimatoprost 0.03% ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost 0.01% ophthalmic solution — One drop of bimatoprost 0.01% ophthalmic solution instilled to each eye, once daily in the evening for 2 years.
  Other Names: LUMIGAN® 0.01%; LUMIGAN 0.1 mg/ml
  Arms: Bimatoprost 0.01% Ophthalmic Solution
Drug: bimatoprost 0.03% ophthalmic solution — One drop of bimatoprost 0.03% ophthalmic solution instilled to each eye, once daily in the evening for 2 years.
  Other Names: LUMIGAN® 0.03%; LUMIGAN 0.3 mg/ml
  Arms: Bimatoprost 0.03% Ophthalmic Solution

SUMMARY:
This study will evaluate the long-term safety of bimatoprost 0.01% ophthalmic solution compared with bimatoprost 0.03% ophthalmic solution in patients with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or glaucoma in each eye
* Requires intraocular pressure (IOP)-lowering therapy in both eyes
* Best corrected visual acuity of 20/100 or better in each eye

Exclusion Criteria:

* Ocular seasonal allergies within 2 years
* Required chronic use of ocular medications during the study (intermittent use of artificial tears is allowed)
* Ocular surgery or laser within 3 months
* Anticipated wearing of contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Hansen, Study Director — Allergan
Locations (50):
- Belgium (2):
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
- Czechia (2):
  - University Hospital Brno, Brno
  - Eye Clinic, Frýdštejn
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Clinique Montcelli, Marseille
- Germany (6):
  - Universitat Augenklinik, Freiburg im Breisgau
  - Univ. des Saarlandes, Homburg Saar
  - Johannes Gutenberg Univ Mainz, Mainz
  - Thelen Private Practice, Műnster
  - Augenzentrum Siegburg, Siegburg
  - Department of Ophthalmology, University of Tuebingen, Tübingen
- Hungary (4):
  - Budapest Retina Associates Kft., Budapest
  - University Med. School of Debrecen, Debrecen
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - University of Szeged Szent-Gyorgyi Albert Clinical Center, Szeged
- Israel (5):
  - Carmel Medical Center, Haifa
  - Glaucoma Service The Rabin Medical Center, Petach Tiqva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - Azienda Ospedaliera Universitaria, Catania
  - Azlenda Ospedaliero Universitaria Careggi Viale, Florence
  - Istituto Scientifico San Raffaele, Milan
  - Dipartimento di Scienze Otorino-Odonto-Oftalmologiche e Cerv, Parma
  - Fondazione G.B. Bietti per l'Oftalmologia I.R.C.C.S., Rome
- Poland (7):
  - EuroMedic Kliniki Specjalistyczne, Katowice
  - ZOZ OKO- TEST Poradnia Okulistyczna, Nowy Targ
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu, Poznan
  - Samodzielny Publiczny Szpital, Szczecin
  - Osrodek Badan Klinicznych Euromedis Sp. z o.o., Szczecin
  - Samodzielny Szpital Kliniczny, Warsaw
  - Akad. Med. w Warszawie - Ketedra I Klin. Okulistki Wyzialu L, Warsaw
- Spain (10):
  - Centro de Ojos de La Coruña, A Coruña
  - Hospital de Torrevieja, Alicante
  - Instituro Condal de Oftalmologia, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - Valles Oftalmologia Recerca, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Instituto oftalmologico Fernandez Vega, Oviedo
  - Fundacion Oftalmologica Del Mediterraneo, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - Birmingham & Midland Eye Center, Birmingham
  - Huntingdon Glaucoma Diagnostic & Research Centre, Huntingdon
  - Western Eye Hospital, London
  - St Thomas' Hospital, London
  - Norfolk and Norwich Hospital, Norwich
  - University Hospital Nottingham, Nottingham
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.01% Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Started | 403 | 403
Safety Population: Received Study Drug | 400 | 398
Completed | 302 | 303
Not Completed | 101 | 100
Not completed — Adverse Event | 50 | 51
Not completed — Lack of Efficacy | 9 | 14
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Protocol Violation | 6 | 4
Not completed — Other Miscellaneous Reasons | 16 | 15
Not completed — Did not Receive Study Drug | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Safety Population, all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.01% Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution | Total
Number analyzed (Participants) | 400 | 398 | 798
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.0) | 62.2 (11.5) | 62.4 (11.3)
Age, Customized [Number; unit: participants]
  < 45 years | 22 | 26 | 48
  ≥ 45 years to ≤ 65 years | 216 | 211 | 427
  > 65 years | 162 | 161 | 323
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 187 | 384
  Male | 203 | 211 | 414

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting One or More Treatment-Related Ocular Surface Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The percentage of participants with ocular (eye) surface AEs deemed related to treatment by the investigator are reported.
Time Frame: 24 Months
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost 0.01% Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 400 | 398
percentage of participants | 33.3 | 37.7
Statistical Analysis 1: Comparison: Bimatoprost 0.01% Ophthalmic Solution vs Bimatoprost 0.03% Ophthalmic Solution; Test type: Superiority or Other; p = 0.148, Cochran-Mantel-Haenszel — P-value was stratified by baseline prostaglandin analogue (PGA) treatment(yes/no) and by baseline active ocular surface finding (present/absent); Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-11 to 1.9] — bimatoprost 0.01% ophthalmic solution - bimatoprost 0.03% ophthalmic solution

2. Secondary Outcome: Percentage of Participants Reporting One or More Treatment-Related Ocular Surface Adverse Events Excluding "Conjunctival Hyperemia"
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The percentage of participants with ocular (eye) surface AEs deemed related to treatment by the investigator excluding AEs with the preferred term Conjunctival hyperemia are reported.
Time Frame: 24 Months
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost 0.01% Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 400 | 398
percentage of participants | 26.0 | 29.6

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Safety Population, all participants who received at least one dose of study drug, was used to determine the number of participants at risk for Serious and Non-serious Adverse Events.
Arm/Group | Bimatoprost 0.01% Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 45/400 | 40/398
Other Adverse Events (participants affected / at risk) | 167/400 | 186/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bimatoprost 0.01% Ophthalmic Solution (N=400) | Bimatoprost 0.03% Ophthalmic Solution (N=398)
Intraocular pressure fluctuation (Investigations) | 4 | 2
Cataract (Eye disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Intraocular pressure increased (Investigations) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Cataract cortical (Eye disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1/197 | 0/187
Vitreous adhesions (Eye disorders) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/203 | 1/211
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Echinococciasis (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Inguinal hernia repair (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Optic neuropathy (Eye disorders) | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% Ophthalmic Solution (N=400) | Bimatoprost 0.03% Ophthalmic Solution (N=398)
Blepharitis (Eye disorders) | 14 | 23
Cataract (Eye disorders) | 20 | 24
Conjunctival hyperaemia (Eye disorders) | 80 | 90
Dry eye (Eye disorders) | 36 | 42
Eye pain (Eye disorders) | 21 | 20
Foreign body sensation in eyes (Eye disorders) | 11 | 21
Punctate keratitis (Eye disorders) | 22 | 30
Influenza (Infections and infestations) | 26 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.